CLINICAL TRIAL: NCT05513807
Title: Graft Acute Kidney Injury: Vitamin B3 to Facilitate Renal Recovery In the Early Life of a Transplant - GABRIEL
Brief Title: Graft Acute Kidney Injury: Vitamin B3 to Facilitate Renal Recovery In the Early Life of a Transplant
Acronym: GABRIEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200036
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Delayed Graft Function
Keywords: Kidney Transplantation; Delayed Graft Function; Niacinamide (NAM); Acute Kidney Injury; Acute Tubular Necrosis; creatinine reduction ratio; Nicotinamide Adenine Dinucleotide; Quinolinate; urinary quinolinate / tryptophane
MeSH Terms: conditions — Delayed Graft Function; Acute Kidney Injury; Kidney Cortex Necrosis | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Experimental)
  Interventions: Drug: Nicotinamide treatment
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo treatment

INTERVENTIONS:
Drug: Nicotinamide treatment — 3g Nicotinamide orally (1g immediately pre transplant, then immediately 1g post-transplant after the recovery room and 1g 24 hours later)
  Other Names: NICOBION
  Arms: Nicotinamide
Drug: Placebo treatment — 3g Placebo orally (1g immediately pre transplant, then immediately 1g post-transplant after the recovery room and 1g 24 hours later)
  Arms: Placebo

SUMMARY:
Delayed graft function occurs in more than 20% of kidney transplantations. It is an episode of post-ischemic acute kidney injury with long-term consequences on the allograft's function. Based on preclinical data and on a stage 1 clinical trial, the hypothesize is that an acquired defect in NAD+ biosynthesis is instrumental in delayed graft function and that a treatment with high doses of vitamin B3 (nicotinamide) will improve the early renal graft function.

Thus, it is planned to recruit 204 kidney allograft recipients immediately before transplantation and randomize them to either placebo or nicotinamide treatment for 3 administrations before transplantation, immediately after it and on the next day.

The efficacy of nicotinamide to foster early graft function will be evaluated by comparing the creatinine reduction ratio between the placebo and the nicotinamide treated groups.

Serum will be collected before and 2 days after transplantation and urine 2 days and 3 months after transplantation to study the relationship between biological markers of NAD+ biosynthesis and nicotinamide's effect on early kidney graft function.

DETAILED DESCRIPTION:
Delayed graft function (DGF) is a frequent event in kidney transplantation (nationwide, 20.9% if all kinds of donors are included), and is prejudicial to graft survival. DGF is mostly due to acute tubular necrosis (ATN), induced by different cycles of renal ischemia (cold and warm). Until now, ATN has no specific treatment. Nicotinamide (NAM), also known as vitamin PP or as a vitamin B3 analog has recently emerged as a major therapeutic option to prevent ATN and accelerate its recovery. NAM actually allows maintaining mitochondrial function in the context of renal ischemia. In humans, NAM given orally (1 and 3g/day for 3 days) was shown to be effective in a phase I study and was associated with a 35% decreased incidence of AKI in 41 high-risk cardiac surgery patients. It has a well-known and highly favorable safety profile.

The GABRIEL study aims at testing its beneficial properties in the specific context of DGF in phase III study. The early kidney allograft function will be assessed on the creatinine reduction ratio between days 1 and 2 (CRR2, calculated by the following formula: CRR2 (%) = ([Cr1-Cr2]×100)/Cr1, where Cr1 and Cr2 are the morning serum creatinine on post-operative day 1 and day 2 respectively.

The objectives are also to :

1. Verify the safety profile of NAM (liver toxicity and tacrolimus trough levels to detect an interaction)
2. Evaluate the effect of NAM on the rate of delayed graft function defined conventionally as the need for dialysis before POD7.
3. Evaluate the effect of NAM on renal graft function 3 months after transplantation.
4. Evaluate the effect of NAM on serum NAM levels (difference between NAM at POD2 and NAM at baseline)
5. Evaluate the effect of NAM on the biopsy-proven rejection rate within three months after transplantation.
6. Measurement accuracy, and positive predictive value of the urinary quinolinate / tryptophane ratio measured early after transplantation (at POD2) for CRR2, DGF, and graft function estimated by MDRD at 3 months.
7. Evaluate the effect of NAM serum concentration at baseline on the level of risk of DGF.
8. Cost-effectiveness of NAM after transplantation of a kidney from a deceased donor.
9. Comparison of different separation techniques (LC, HILIC, IC, EC) for MS quantification of uQ/T and serum NAM.

Patients called for transplantation will be included if they meet the required criteria. After inclusion and according to randomization, the patient will receive the first dose of treatment (1g NAM or placebo, V0) immediately before surgery, at the time of induction of immunosuppression. The second dose will be given to the patient immediately after recovery room (POD1), and the third dose 24 hours thereafter (POD2). NAM administrations will be no less than 8 and no more than 26 hours apart. The biological samples and anamnestic items will be collected between 6 and 10 AM on the prespecified visits.

A quality of life questionnaire EQ5D will be completed by the patient at V0 after inclusion and before transplantation ; and others EQ5D questionnaires will be completed at POD7 and last study visit M3.

It is expected that this study will inform on the effect of NAM on early graft function, and help to define its potential place in the management of a subset if not all kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years,
* Patients in end stage renal disease (ESRD) requiring dialysis (hemodialysis or peritoneal dialysis),
* Kidney transplant with deceased donor (brain death or cardiac death Maastricht 3),
* Affiliation to French social security ("AME" excepted),
* Written informed consent

Exclusion Criteria:

* Preemptive transplant,
* Pregnancy,
* Liver disease defined by the necessity for a specialized follow-up by an hepatologist (with liver biological results disturbed) or by elevated liver enzymes > 3N (ALAT and/or gammaGT) on the day of transplantation
* Transplantation of multiple organs,
* Hypersensitivity to nicotinamide or one of excipients,
* Participation to another interventional study (RIPH1),
* Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Efficacy of 3 doses of NAM given orally at 1g/dose immediately pre transplant and during the first 2 post-operative days of renal transplantation versus placebo, on the early graft function, assessed by CRR2. | Post-Operative Day 2
  The primary endpoint is based on creatinine reduction ratio between days 1 and 2 (CRR2, calculated by the following formula: CRR2 (%) = ([Cr1-Cr2]×100)/Cr1, where Cr1 and Cr2 are the morning serum creatinine on post-operative day 1 and day 2 respectively.

SECONDARY OUTCOMES:
Verify the safety profile of NAM (liver toxicity and tacrolimus trough levels to detect an interaction) | Post-Operative Day 7
  Proportion of patients with at least one increase of ALAT concentrations > 2N between V0 and POD7 (mild and reversible liver toxicity has been described with high dose NAM treatment ; and proportion of patients with inadequately high tacrolimus trough levels (> 20 ng/mL) at POD2, and POD7.
Evaluate the effect of NAM on the rate of delayed graft function defined conventionally as the need for dialysis before POD7 | Post-Operative Day 7
  Rate of DGF (Delayed Graft Function), as defined by the need of at least one dialysis between engraftment and POD7
Evaluate the effect of NAM on renal graft function 3 months after transplantation | 3 months after transplantation
  Correlation between CRR2 and :
  1. eGFR 3 months after transplantation among patients with no renal event such as, rejection, pyelonephritis and obstruction.
  2. Urinary quinolinate/tryptophan ratio measured by mass spectrometry at 3 months after transplantation among patients with no renal event such as, rejection, pyelonephritis and obstruction
Evaluate the effect of NAM on serum NAM levels (difference between NAM at POD2 and NAM at baseline) | Post-Operative Day 2
  Comparison of NAM concentration variation from baseline to POD2.
Evaluate the effect of NAM on the biopsy-proven rejection rate within three months after transplantation. | 3 months after transplantation
  Proportion of patients with at least one episode of biopsy-proven rejection (T-cell or antibody mediated) as per the Banff's 2017 classification criteria (48) within 3 months after transplantation
Measurement accuracy, and positive predictive value of the urinary quinolinate / tryptophane ratio measured early after transplantation (at POD2) for CRR2, DGF, and graft function estimated by MDRD at 3 months | Post-operative Day 2
  Urinary quinolinate/tryptophan ratio measured by mass spectrometry at POD2 where we expect an increase in patients with DGF and also at M3, to determine the reversibility of the metabolic abnormalities.
Evaluate the effect of NAM serum concentration at baseline on the level of risk of DGF | 3 months after transplantation
  Serum concentration of NAM at baseline (before pre transplant NAM dose), measured by mass spectrometry
Cost-effectiveness and cost utility of NAM after transplantation of a kidney from a deceased donor | Baseline
  Incremental cost effectiveness ratio of NAM compared to placebo, measured by the difference in costs of healthcare divided by the difference in rate of 3-month renal events defined as rejection, pyelonephritis and obstruction and incremental cost utility analysis using quality adjusted life years
Comparison of different separation techniques (LC, HILIC, IC, EC) for MS quantification of uQ/T and serum NAM | Baseline, POD2 and 3 months after transplantation
  Reproductibility of the quantification of urinary quinolinate/tryptophan ratio and serum concentration of NAM, measured by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Pierre GALICHON, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Renal Transplantation - Hospital Pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Biological samples collection :
  During the study, serum at V0 and POD2, and urine at POD2 and M3 will be aliquoted into three, and stored at -80°C or -20°C. Aliquots will be sent in dry ice to the Biological Resource Center at Pitié-Salpêtrière Hospital (CRB-PSL).
  * 1 aliquot of each visit (baseline, POD2 and M3) will be send for analysis for the study
  * The last aliquots will be sent to UMRS1155-INSERM - Maladies Rénales Fréquentes et Rares : des Mécanismes Moléculaires à la Médecine Personnalisée (4 rue de la Chine 75020 Paris) where all study samples will be centrally stored at -80°C under the supervision of Pr. Pierre Galichon in a biological sample collection for further analysis which may be useful for investigation of renal graft functional recovery in light of advances in scientific knowledge, provided the participant is informed and does not oppose this, as stated in the information note/consent form. The total period of conservation couldn't exceed 5 years.